CLINICAL TRIAL: NCT01206101
Title: A 52 Week Randomized, Double-Blind, Placebo Controlled, Parallel Group, Multi-Center, Multinational Trial In Islet Cell Transplant Subjects With Type 1 Diabetes Mellitus To Determine If The Early Use Of Liraglutide As An Adjunct To Standard Care Increases The Proportion Of Subjects Achieving Insulin Independence After First Transplantation
Brief Title: Efficacy and Safety of Liraglutide in Subjects With Type 1 Diabetes Undergoing Islet Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision to close the NN2211-3619 trial was based on the very low recruitment rate as well as challenges relating to trial execution and study completion.
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-3619; 2009-013090-18 (EudraCT Number); U1111-1114-8952 (Other: WHO)
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- Liraglutide placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Dose escalation of liraglutide up to 1.2 to 1.8 mg before islet cell transplant until the planned number of transplanted subjects is complete or subject is transplanted. After islet cell transplant, subjects continue to receive the reached liraglutide dose for 52 weeks. Injected subcutaneously(under the skin) once daily.
  Arms: Liraglutide
Drug: placebo — Dose escalation escalation of liraglutide up to 1.2 to 1.8 mg before islet cell transplant until the planned number of transplanted subjects is complete or subject is transplanted. After islet cell transplant, subjects continue to receive the reached liraglutide placebo dose for 52 weeks. Injected subcutaneously (under the skin) once daily.

SUMMARY:
This trial is conducted in Europe and North America. The aim of this trial is to investigate if liraglutide treatment can increase the proportion of insulin-independent subjects one year after islet cell transplantation who required only one (single-donor) islet cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least 5 years
* Candidate for islet cell transplantation based upon local accepted practice and guidelines
* Reduced awareness of hypoglycaemia

Exclusion Criteria:

* Treatment with any anti-diabetic medication other than insulin including insulin pump within 4 weeks of trial start
* Any previous organ transplantation
* A history of acute idiopathic or chronic pancreatitis
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-03-21 (Actual); Primary Completion 2013-06-03 (Actual); Study Completion 2013-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (16):
- United States (4):
  - Novo Nordisk Investigational Site, Duarte, California
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Madison, Wisconsin
- Canada (2):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
- France (5):
  - Novo Nordisk Investigational Site, Besançon
  - Novo Nordisk Investigational Site, Grenoble
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Strasbourg
- Novo Nordisk Investigational Site, Dresden, Germany
- Switzerland (2):
  - Novo Nordisk Investigational Site, Geneva
  - Novo Nordisk Investigational Site, Zurich
- United Kingdom (2):
  - Novo Nordisk Investigational Site, Headington
  - Novo Nordisk Investigational Site, London

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 3 sites in 3 countries:
  Canada: 1 site; Switzerland: 1 site; US: 1 site.
Pre-assignment Details: All the subjects were on pre-trial insulin at screening.
Groups:
- Liraglutide: Liraglutide was injected subcutaneously once-daily. The dose of liraglutide was escalated up to 1.8 mg (or 1.2 mg if 1.8 mg not tolerated) prior to islet cell transplant and continued until one year after the first transplant in each subject.
- Liraglutide Placebo: Liraglutide placebo was injected subcutaneously once-daily. The dose of liraglutide placebo was escalated up to 1.8 mg (or 1.2 mg if 1.8 mg not tolerated) prior to islet cell transplant and continued until one year after the first transplant in each subject.
Period: Overall Study
Arm/Group | Liraglutide | Liraglutide Placebo
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Unclassified | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Liraglutide Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion Of Insulin-independent Subjects After Receiving Only One (Single-Donor) Islet Cell Transplant
Description: Proportion Of Insulin-independent Subjects After Receiving Only One (Single-Donor) Islet Cell Transplant.
Time Frame: At week 52 after initial transplantation
Population: Full analysis set (FAS) - all randomised subjects who underwent one or more transplantations after randomisation. Due to the premature termination of the trial prior to islet cell transplantation in any randomised subject, no formal statistical analyses were performed.
Arm/Group | Liraglutide | Liraglutide Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: A hypoglycaemic episode was defined as treatment emergent if the onset of the episode was on or after the first day of exposure to randomised treatment and until the last day on randomised treatment. Confirmed hypoglycaemic episodes were categorised either as minor (PG<3.1 mmol/L [56 mg/dL]) or severe (subject unable to treat himself/herself).
Time Frame: During week 0 to week 52
Population: as for outcome 1
Arm/Group | Liraglutide | Liraglutide Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Proportion of Subjects With HbA1c Below Or Equal to 6.5% At Week 52 That Are Free From Severe Hypoglycaemic Events
Description: Proportion of subjects with HbA1c below or equal to 6.5% at week 52 that were free from severe hypoglycaemic events
Time Frame: From week 0 to week 52 after initial transplantation
Population: as for outcome 1
Arm/Group | Liraglutide | Liraglutide Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Proportion of Insulin-Independent Subjects
Description: Proportion of insulin-independent subjects among all randomised subjects who had one or more transplantations after randomisation
Time Frame: At 52 weeks after initial transplantation
Population: as for outcome 1
Arm/Group | Liraglutide | Liraglutide Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Islet Cell Yield During Culture
Description: Change in islet cell yield from pre-culture to post-culture
Time Frame: From 0 hours pre-culture to 24 hours to 72 hours
Population: as for outcome 1
Arm/Group | Liraglutide | Liraglutide Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Glucose Level Variability And Hypoglycaemia Duration Derived From The Continuous Glucose Monitoring System (CGMS)
Description: Change from baseline in glucose level variability and hypoglycaemia at baseline, weekly during liraglutide dose escalation, at 12 weeks pre-transplant, at 24 weeks post-transplant, 52 weeks post-transplant and 56 weeks (4 weeks after withdrawal of liraglutide or liraglutide placebo)
Time Frame: At 12 weeks pre-transplant, at 24 weeks post-transplant, 52 weeks post-transplant and 56 weeks (4 weeks after withdrawal of liraglutide or liraglutide placebo)
Population: as for outcome 1
Arm/Group | Liraglutide | Liraglutide Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from week 0 to week 52.
Description: Safety analysis set includes all subjects who received at least one dose of the trial product or its comparator.
Arm/Group | Liraglutide | Liraglutide Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=2) | Liraglutide Placebo (N=1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Computerised tomogram abnormal (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the premature termination of the trial prior to islet cell transplantation in any randomised subject, no results are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.